CLINICAL TRIAL: NCT05234450
Title: Multi-omics Characterization of Pancreatic Neuroendocrine Tumors and Carcinomas
Acronym: Camune
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7561
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Cancer of Pancreas
Keywords: Cancer of Pancreas; Neuroendocrine Tumors; Carcinoma; Neuroendocrine
MeSH Terms: conditions — Pancreatic Neoplasms; Neuroendocrine Tumors; Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this work, the investigators count through the integrated multi-omics analysis to identify different tumor subgroups in pancreatic neuroendocrine tumors and carcinomas regardless of their grade and stage. To achieve this, they will resort to the use of next-generation sequencing approaches (RNAseq, then use of MCP Counter for the absolute quantification of the eight populations of immune cells in the tumor microenvironment), alterations in epigenetics with study of the methylome by MeDIP, ChIPseq, telomere (ALT) study, as well as correlation with peripheral blood neutrophil to lymphocyte ratio and immunohistochemistry data such as Ki67, p53, Rb, DAXX, ATRX, PDL1, immune cell labeling. This will be done on frozen or paraffin material. This work will provide a more complete biological picture of pancreatic neuroendocrine tumors and carcinomas.

ELIGIBILITY:
Inclusion criteria:

* Adult patient (≥18 years old)
* Subject with histologically confirmed tumor or neuroendocrine carcinoma of the pancreas
* Subject with tumors or neuroendocrine carcinoma of the pancreas regardless of the stage of the disease
* Supported at the University Hospitals of Strasbourg between 01/01/2008 and 01/09/2019
* Near therapeutic blood count available (less than 6 months)
* Availability of frozen and/or paraffin tumor material
* Patients who have already given their consent for their biological resources to be kept at the CRB or in the anatomopathology department of the HUS, and subsequently reused, as well as the anonymous data associated with them, for scientific research purposes.

Exclusion criteria:

* Opposition of the patient to participate in the study
* Diagnosis other than pancreatic neuroendocrine tumor
* Biological tissue from a patient who does not meet all the inclusion criteria
* Impossibility of giving informed information to the subject
* Patient under judicial protection En savoir plus sur ce texte sourceVous devez indiquer le texte source pour obtenir des informations supplémentaires Envoyer des commentaires Panneaux latéraux

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) with histologically confirmed tumor or neuroendocrine carcinoma of the pancreas
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Establishment of the number of tumor subgroups by integrating data from all multi-omics analyses | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MALOUF, MD, PhD, Principal Investigator — Service d'Oncologie - CHU de Strasbourg - France
Locations (1):
- Service d'Oncologie - CHU de Strasbourg - France, Strasbourg, France